CLINICAL TRIAL: NCT07178704
Title: PILOT STUDY: The Metabolic and Genetic Drivers of Body Composition Changes Following Weight Loss Surgery
Brief Title: The Metabolic and Genetic Drivers of Body Composition Changes Following Weight Loss Surgery
Status: Recruiting | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 24-0361
Record Dates: First submitted 2025-08-22; First posted 2025-09-17 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Bariatric Surgery Patients
Keywords: Body composition; Sarcopenia; Weight loss surgery; Muscle function; Protein metabolism
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine; Fecal; Plasma; Serum; Foregut tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bariatric Surgery Patients: Patients due to undergo either sleeve gastrectomy or gastric bypass surgery.
- Healthy Control Subjects: Healthy weight individuals recruited from the local population.

SUMMARY:
Weight loss surgery is very good at reducing body weight but it can also cause the loss of both muscle and strength. Some patients undergoing weight loss surgery do not achieve their weight loss goals and regain the weight they lost. When this occurs, the loss of muscle and strength combined with the regain of weight can impact the individual's quality of life and ability to remain active and mobile.

The purpose of this study is to understand the behavioral, biological, and genetic factors that influence the success of weight loss surgery and its impact on muscle mass.

Bariatric surgery patients participating in the trial will be monitored prior to, and for a year following weight loss surgery, with data collected about their eating habits, hand grip strength, and the loss of fat, muscle, and body weight following surgery. Some patients will be additionally invited to undergo detailed metabolic assessment, where we will measure how their body uses nutrients it consumes, the composition of their body (e.g. how much lean and fat tissue they have and where it is stored), identify the bacteria living in their gut, and determine their physical performance. In all patients a small sample of gut tissue will be collected at a routine endoscopy performed in advance of weight loss surgery to identify the expression (activity) of genes in their DNA.

Healthy subjects will also be recruited to allow us to compare between healthy weight individuals and those undergoing weight loss surgery. On a single occasion, the healthy volunteers will undergo the same detailed metabolic assessment performed in patients as described above. We will not examine the bacteria living in the gut of the healthy volunteers, nor will we collect gut tissue from these individuals.

ELIGIBILITY:
Inclusion Criteria (Healthy Volunteers):

* Age: 30 to 50 years at time of consent
* BMI: 20-25 kg.m-2
* Male or Female
* All races and ethnic backgrounds
* Ability to speak and read English
* Subject has provided informed consent in a manner approved by the IRB and is willing and able to comply with the trial procedures.

Inclusion Criteria (Bariatric Surgery Patients):

* Age: 18 to 65 years at time of consent
* BMI: 35-50 kg.m-2
* Scheduled to undergo bariatric surgery at UTMB
* All races and ethnic backgrounds
* Ability to speak and read English
* Subject has provided informed consent in a manner approved by the IRB and is willing and able to comply with the trial procedures.

Additional inclusion criteria for patients undergoing enhanced metabolic assessment:

* Age: restricted to 30 to 50 years of age
* Undergoing gastric bypass surgery

Exclusion Criteria (Healthy Volunteers):

* Heart, vascular, or pulmonary disease
* Uncontrolled blood pressure (systolic BP > 170, diastolic BP > 95 mmHg)
* Impaired renal function (creatinine > 1.5 mg/dl)
* Anemia (hematocrit < 33 % or donated blood in the past 12 weeks.)
* Diabetes mellitus or other untreated endocrine or metabolic disorder
* Recent (5 years or less) history of cancer
* Systemic steroids, anabolic steroids, growth hormone, or immunosuppressant use within 6 months.
* Recent (6 months) adherence to a weight-loss or weight-gain diet, resulting in a weight change of 10% or more.
* Body mass index > 25.5 kg.m-2
* Body mass index < 19.5 kg.m-2 or recent history (< 12 months) of disordered eating.
* Acute infectious disease or chronic infection.
* Pregnancy or breast-feeding.
* Recent (1 month) consumption of protein-based sports supplements.
* Any medical condition that, in the opinion of the investigator, would place the subject at increased risk for participation.
* Known allergic reaction to any agent under investigation or required by the protocol, including Phenylketonuria.
* Unable to lie still in a supine position for 10 minutes.
* History of prior non-compliance or the presence or history of a psychiatric condition (including drug or alcohol addiction) that would, in the opinion of the investigator, make it difficult for the subject to comply with the study procedures or follow the investigators instructions.
* Concurrent participation in another research study.
* Use of an investigational agent in the 30 days prior to signing informed consent.

Exclusion Criteria (Bariatric Surgery Patients):

* Fails the medical criteria for bariatric surgery.
* Anemia (hematocrit < 33 % or donated blood in the past 12 weeks.)
* Recent (5 years or less) history of cancer
* Systemic steroids, anabolic steroids, growth hormone, or immunosuppressant use within 6 months.
* Body mass index < 35 or > 50 kg.m-2.
* Acute infectious disease or chronic infection.
* Pregnancy or breast-feeding.
* Any medical condition that, in the opinion of the investigator, would place the subject at increased risk for participation.
* History of prior non-compliance that would, in the opinion of the investigator, make it difficult for the subject to comply with the study procedures or follow the investigator's instructions.
* Concurrent participation in another research study.
* Use of an investigational agent in the 30 days prior to signing informed consent.

Additional exclusion criteria for patients undergoing enhanced metabolic assessment:

* Known allergic reaction to any agent under investigation or required by the protocol, including Phenylketonuria.
* Unable to lie still in a supine position for 10 minutes.
* Previous bariatric surgery or undergoing a procedure other than gastric bypass (e.g. sleeve gastrectomy).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from those electing to undergo bariatric surgery at the University of Texas Medical Branch. Healthy volunteers will be recruited from individuals responding to adverts targeting the Houston - Galveston region.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Whole-body Protein Turnover Rates | Measured at baseline in both healthy volunteers & patients undergoing metabolic assessment. The latter will undergo repeat assessment on two further occasions across a 1 year period post surgery.
  Whole-body protein turnover rates measured over a 48 hour period, accomplished via the consumption of a drink containing isotopically labelled (15N) alanine and the subsequent collection of urine for two days. Will be performed on a single occasion in healthy volunteers and up to three times in bariatric patients undergoing metabolic assessment.
Association between foregut gene expression and degree of weight reduction | A single occasion from tissue collected during the routine pre-operative upper endoscopy. (baseline)
  Assessed only in patients. Gene expression of the foregut will be analyzed in tissue collected from patients during the routine pre-operative upper endoscopy. Subsequently, participants will be stratified into those achieving: <10%, 10-20%, or >20% weight loss 12 months post-surgery, and differentially expressed genes between the three groups determined.

SECONDARY OUTCOMES:
Dietary Protein Intake | Measured at baseline in both healthy volunteers & patients undergoing metabolic assessment. The latter will undergo repeat assessment on two further occasions across a 1 year period post surgery.
  Dietary protein intake will be determined by participants completing three-day food diaries. This will be performed on a single occasion in healthy volunteers and up to three occasions in bariatric patients undergoing metabolic assessment.
Body weight | Measured at baseline in both healthy volunteers & bariatric surgery patients. The latter will undergo repeat assessment on two further occasions across a 1 year period post surgery.
  Body weight will be determined using digital scales (in kg). Procedures will be performed on a single occasion in healthy volunteers and up to three times in bariatric patients.
Body composition | Measured at baseline in both healthy volunteers & bariatric surgery patients undergoing metabolic assessment. The latter will undergo repeat assessment on two further occasions across a 1 year period post surgery.
  Body composition will be determined in patients by whole-body bioelectrical impedance. Regional body composition will be additionally assessed in healthy volunteers and bariatric surgery patients undergoing metabolic assessment via whole-body dual-energy x-ray absorptiometry (DXA) imaging. Procedures will be performed on a single occasion in healthy volunteers and up to three times in bariatric patients undergoing metabolic assessment.
Short Physical Performance Battery Test | Measured at baseline in both healthy volunteers & bariatric surgery patients. The latter will undergo repeat assessment on two further occasions across a 1 year period post surgery.
  Assessed using the established short physical performance battery (SPPB) test. Will be performed on a single occasion in healthy volunteers and up to three times in bariatric patients undergoing metabolic assessment.
Handgrip Strength | Measured at baseline in both healthy volunteers & bariatric surgery patients. The latter will undergo repeat assessment on two further occasions across a 1 year period post surgery.
  Assessed using a handgrip dynamometer (in kg). Will be performed on a single occasion in healthy volunteers and up to three times in bariatric patients.
Physical Activity levels (accelerometry) | Measured at baseline in both healthy volunteers & bariatric surgery patients. The latter will undergo repeat assessment on two further occasions across a 1 year period post surgery.
  Assessed by having individuals wear an accelerometer for up to 7 days, allowing step counts and energy expenditure to be determined. Will be performed on a single occasion in healthy volunteers and up to three times in bariatric patients undergoing metabolic assessment.
Energy Intake | Measured at baseline in both healthy volunteers & bariatric surgery patients undergoing metabolic assessment. The latter will undergo repeat assessment on two further occasions across a 1 year period post surgery.
  Energy intake assessed via the completion of a 3-day food diary. Will be performed on a single occasion in healthy volunteers and up to three times in bariatric patients undergoing metabolic assessment.
Energy Expenditure | Measured at baseline in both healthy volunteers & bariatric surgery patients undergoing metabolic assessment. The latter will undergo repeat assessment on two further occasions across a 1 year period post surgery.
  Energy expenditure will be determined at rest via indirect calorimetry. Will be performed on a single occasion in healthy volunteers and up to three times in bariatric patients undergoing metabolic assessment.

OTHER OUTCOMES:
Changes in the Gut Microbiome post-bariatric surgery | Measured at baseline and two further occasions across a 1 year period post surgery.
  (Measured in patients undergoing metabolic assessment only). The gut microbiome will be analyzed in fecal samples collected from patients, with the type and number of bacteria colonizing the gut determined using established RNA sequencing approaches. Significant changes in the colonizing bacteria in response to surgery will be determined via the collection of samples before surgery (baseline) and two further occasions over a 1 year period following bariatric surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Murton, PhD, Principal Investigator — The University of Texas Medical Branch
Locations (1):
- The University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Given the small participant numbers involved, the sharing of individual participant data could carry the risk of re-identification of the study participants, despite the data being provided in de-identified form.